CLINICAL TRIAL: NCT06850649
Title: Investigation of the Clinical Outcomes of Endocrowns Manufactured From Three Different Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulcan COSKUN AKAR (Other)
Responsible Party: Sponsor-Investigator, Gulcan COSKUN AKAR, Ege University Scientific Research Project, Ege University
Organization: Ege University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-61749811-000-1963653
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gross Material Loss in Endodontically Treated Upper and Lower Molars; No Systemic Infection; Gingival Steps Should be at Gum Level
Keywords: endodontic treatment; CAD-CAM; endocrown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endocrown Materials (Experimental): IPS Empress CAD Vita Enamic VarseoSmile Crown Plus
  Interventions: Other: endocrowns

INTERVENTIONS:
Other: endocrowns — IPS Empress CAD Vita Enamic VarseoSmile Crown Plus

SUMMARY:
The goal of this clinical trial is to examine the durability of endocrowns, created using various materials and manufacturing techniques with a fully digital workflow, and their ability to maintain functionality and aesthetics in the oral cavity.

The main questions it aims to answer were does effect of different materials on clinical success?

DETAILED DESCRIPTION:
Based on the power analysis, it was determined that restorations would be applied to 11 teeth in each of the three material groups (lithium-disilicate reinforced glass-ceramic, polymer infiltrated ceramic, and 3D-printed permanent hybrid resin) as well as the control group (n=11). A total of 33 teeth received endocrown restorations. Additionally, 11 patients were directly restored with composite resin in molar teeth with MOD cavities.

The digital impressions of the patients receiving endocrown restorations were recorded using an intraoral optical scanner and sent to a specialized dental laboratory. For two of the groups (lithium disilicate-reinforced glass-ceramic, polymer infiltrated ceramic), restorations were fabricated using block milling, while for the third group (permanent hybrid resin), restorations were produced through 3D printing. The restorations were cemented adhesively. The restorations were evaluated using the Modified FDI and Modified USPHS criteria at baseline (0) and at the 6-month follow-up, and the data were subjected to statistical analysis.

At the 6-month evaluation, a statistically significant difference in color match was found between the groups based on the Modified FDI criteria, whereas no statistically significant differences were observed for any of the Modified USPHS criteria. All endocrowns produced with the three different materials survived and showed clinical success at the 6-month follow-up. Nevertheless, additional clinical studies with extended follow-up durations are required.

ELIGIBILITY:
Inclusion Criteria:

* Must be a lower or upper molar tooth
* Must be periodontal healthy
* There must be at least two axial walls in the relevant tooth
* Gingival steps should be at gum level
* There must be neighboring teeth mesial and distal to the relevant tooth.
* The place where it occludes must be the opposing tooth and the tooth must be a natural or filled tooth without a prosthesis.
* No systemic acut or chronic conditions (Thyroid disease, Alzheimer's Disease, Insulin dependent diabetes, etc.)

Exclusion Criteria:

* Inadequate oral hygiene, bleeding on probing, pocket deeper than 3 mm mobility presence
* Sensitivity to percussion after root canal treatment
* Insufficient enamel tissue remaining in the relevant tooth
* Presence of radiographically abnormal periodontal space
* Teeth with inadequate bone support
* Teeth with root resorption and fracture

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes | 6 month
  Restorations were checked clinically at the time of delivery and 6 months later. A 0.15 mm probe (DEPPELER 150EX, Rolle, Switzerland) was used for the controls.
  Modified USPHS and modified FDI criteria (revised 2023) were used in the evaluations.
  The modified USPHS criteria were recorded as Alpha (A), Bravo (B), Charlie (C), Delta (D), and the modified FDI criteria were recorded as very good, good, adequate, unsatisfactory, and failed.
  'Surface Luster, Surface and Marginal Staining, Colour match and Translucency, Esthetic Anatomical Form, Fracture Material and Retention, Marginal adaptation as Modified FDI Criteria and Marginal Discoloration, Marginal Integrity, Surface Texture, Wear, Postoperative Sensitivity and Recurrent Caries as Modified USPS Criteria were evaluated.
  In the study, the headings of the result measurement tables will be created as follows:
  Comparison of Baseline Modified USPHS Values According to Groups Comparison of Baseline Modified FDI Values According to G

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No